CLINICAL TRIAL: NCT05504213
Title: A Phase Ib, Open-label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of HS-10352 in Combination With Fulvestrant in Patients With Hormone Receptor (HR) Positive, Human Epidermal Growth Factor 2 (HER2)-Negative, PIK3CA Mutation, Locally Advanced or Metastatic Breast Cancer
Brief Title: A Phase Ib Study of HS-10352 Plus Fulvestrant in Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10352-102
Record Dates: First submitted 2022-05-17; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: dose-escalation; dose-expansion; advanced breast cancer; hormone receptor positive; PIK3CA gene mutation
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Endocrine therapy-resistant (Stage 1) (Experimental): Participants who are endocrine therapy pre-treated will be administrated at escalating doses orally of HS-10352 in combination with fulvestrant (500 mg, intramuscular).
  Interventions: Drug: HS-10352 combined with fulvestrant (Stage 1)
- Cohort 2: Endocrine therapy-resistant (Stage 2) (Experimental): Participants who are endocrine therapy-resistant will be treated with HS-10352 orally at the MTD/MAD identified in Stage 1 or/and lower dose in combination with fulvestrant (500 mg, intramuscular)
  Interventions: Drug: HS-10352 combined with fulvestrant (Stage 2)
- Cohort 3: Endocrine therapy-sensitive or endocrine-naïve (Stage 2) (Experimental): Participants who are endocrine therapy-sensitive or naïve will be treated with HS-10352 orally at MTD/MAD or/and lower dose identified in Stage 1 in combination with fulvestrant (500 mg, intramuscular)
  Interventions: Drug: HS-10352 combined with fulvestrant (Stage 2)

INTERVENTIONS:
Drug: HS-10352 combined with fulvestrant (Stage 1) — Drug: HS-10352 HS-10352 will be administered at escalating doses orally once daily on a continuous dosing schedule starting on Cycle 1 Day 1 (C1D1) in a 28 day cycle.
  Drug: Fulvestrant Fulvestrant is administered at a dose of 500 mg intramuscular on Cycle 1 Day 1, Day 15, and Day 1 of every cycle thereafter (where a cycle is 28 days).
  Arms: Cohort 1: Endocrine therapy-resistant (Stage 1)
Drug: HS-10352 combined with fulvestrant (Stage 2) — Drug: HS-10352 participants will be enrolled into Cohort 2 (endocrine therapy-resistant) and Cohort 3 (endocrine therapy-sensitive or naïve) respectively and HS-10352 will be administered at the recommended dose identified in Part 1.
  Drug: Fulvestrant Fulvestrant is administered at a dose of 500 mg intramuscular on Cycle 1 Day 1, Day 15, and Day 1 of every cycle thereafter (where a cycle is 28 days).
  Arms: Cohort 2: Endocrine therapy-resistant (Stage 2); Cohort 3: Endocrine therapy-sensitive or endocrine-naïve (Stage 2)

SUMMARY:
HS-10352 is a highly potent and selective small molecule inhibitor of phosphoinositide 3-kinase (p110α). The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK), and efficacy of HS-10352 plus fulvestrant in patients with hormone receptor (HR) positive, human epidermal growth factor 2 (HER2)-negative, advanced breast cancer (ABC) harboring PIK3CA mutations.

DETAILED DESCRIPTION:
This is a Phase Ib open-label, 2-Part, multi-center study in China. The study will be conducted in two stages: Stage 1 is the dose-escalation part, which is designed to evaluate the safety, tolerability, PK and efficacy, as well as to determine the maximum tolerable dosage (MTD) or maximum applicable dose (MAD) of HS-10352 in combination with fulvestrant. Stage 2 is the dose-expansion part, which is aimed to further assess the efficacy, safety, tolerability and PK, and to establish the recommended phase 2 dose (RP2D) of HS-10352 in combination with fulvestrant.

All participants will be carefully monitored for adverse events (AE) during the study treatment and for 28 days after the last dose of study drug. The PK characteristics of HS-10352 and fulvestrant will be evaluated from C1 to C6. Subjects of this study will be assessed for progression once every 8 weeks until objective disease progression or withdrawal from the trial. As the disease progresses, survival follow-up is recommended bimonthly.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years
2. HR+ HER2- breast cancer confirmed by histology or cytology.
3. Locally advanced disease not amenable to curative treatment by surgery or metastatic disease.
4. Have adequate tumor tissue for the analysis of PIK3CA mutational status. At dose expansion stage, participants should be identified as PIK3CA-mutation positive before enrollment.
5. Females should have postmenopausal status due to either surgical/natural menopause or ovarian suppression with a luteinizing hormone releasing hormone (LHRH) agonist before enrollment. Males should be pre-treated with a LHRH agonist.
6. Have either measurable disease per RECIST v1.1 criteria or at least one predominantly lytic bone lesion must be present.
7. ECOG performance status was 0-1 and did not deteriorate in the previous 2 weeks.
8. Estimated life expectancy for at least three months
9. Females should be using adequate contraceptive measures and should not be breastfeeding at the time of screening, during the study and until 6 months after completion of the study; and have negative results of blood pregnancy test prior to C1D1.

   Males should be using adequate contraceptive measures at the time of screening, during the study and until 6 months after completion of the study.
10. Have signed Informed Consent Form
11. Dose escalation stage-Cohort 1: subjects resistant to endocrine therapy Dose expansion stage-Cohort 2: subjects resistant to endocrine therapy Dose expansion stage-Cohort 3: endocrine therapy-sensitive or endocrine-naive subjects

Exclusion Criteria:

1. Participant with symptomatic visceral disease or any disease burden that makes the participant ineligible for endocrine therapy per the investigator's best judgment
2. Treatment with any of the following:

   1. Previous or current treatment with PI3K, AKT or mTOR inhibitors
   2. For expansion stage, prior treatment with fulvestrant
   3. Any cytotoxic chemotherapy, investigational agents within 21 days of the first dose of study drug; anticancer drugs which have been received within 14 days before the first administration.
   4. Radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study drug, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks of the first dose.
   5. Major surgery (including craniotomy, thoracotomy, or laparotomy, etc.) within 4 weeks of the first dose of study drug.
3. With inflammatory breast cancer at screening.
4. Inadequate bone marrow reserve or organ function.
5. Uncontrolled pleural effusion or ascites or pericardial effusion.
6. Known and untreated, or active central nervous system metastases.
7. History of primary or secondary diabetes.
8. History of acute or chronic pancreatitis
9. Refractory nausea, vomiting, or chronic gastrointestinal diseases, or inability to swallow the study drug that would preclude adequate absorption of HS-10352 or fulvestrant.
10. History of hypersensitivity to any active or inactive ingredient of HS-10352/ fulvestrant or to drugs with a similar chemical structure or class to HS-10352.
11. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
12. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
[Stage 1] Maximum tolerated dose (MTD) of HS-10352 in combination with fulvestrant | Cycle 1 (28 days)
  MTD is defined as the previous dose level at which 2 or more out of 2~6 subjects experienced a DLT.
[Stage 1] Maximum applicable dose (MAD) of HS-10352 in combination with fulvestrant | Cycle 1 (28 days)
  MAD is defined as follows: a) based on PK data, it is anticipated that at this dose level, the dose-exposure plateau has been reached, b) based on existing safety data, it is judged that dose escalation following this dose level will have a large safety risk or subject intolerance, or c) based on the PK-PD model, it suggested that the optimal target concentration of safety and efficacy has been explored.
[Stage 2] Objective response rate (ORR) of HS-10352 in combination with fulvestrant | From the date of first dose until the date of disease progression or withdrawal from study, approximately 3 years
  ORR is defined as the proportion of participants with best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) based on assessment per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
[Stage 1 and Stage 2] Incidence and severity of treatment-emergent adverse events | From Cycle 1 Day 1 (C1D1) until 28 days after the final dose. A cycle is 28 days.
  Assessed by number and severity of adverse events as evaluated according to NCI CTCAE v5.0.
[Stage 1 and Stage 2] PK parameters: the maximum concentration (Cmax) of HS-10352 | Cycle 1 Day 1 (C1D1)，at the first day of Cycle 1 (each cycle is 28 days)
  Defines as the maximum plasma drug concentration of HS-10352
[Stage 1] PK parameters: the maximum concentration (Cmax) of fulvestrant | Cycle 1 (28 days)
  Defines as the maximum plasma drug concentration of fulvestrant
[Stage 1 and Stage 2] PK parameters: time of the maximum concentration (Tmax) of HS-10352 | Cycle 1 Day 1 (C1D1)，at the first day of Cycle 1 (each cycle is 28 days)
  Defined as the time to reach maximum plasma concentration following drug administration of HS-10352
[Stage 1] PK parameters: time of the maximum concentration (Tmax) of fulvestrant | Cycle 1 (28 days)
  Defined as the time to reach maximum plasma concentration following drug administration of fulvestrant
[Stage 1 and Stage 2] PK parameters: elimination half life (t1/2) of HS-10352 | Cycle 1 Day 1 (C1D1)，at the first day of Cycle 1 (each cycle is 28 days)
  Defines as the time measured for the concentration to decrease by one half.
[Stage 1 and Stage 2] PK parameters: area under the concentration-time curve over 24 hours (AUC0-24) of HS-10352 | Cycle 1 Day 1 (C1D1)，at the first day of Cycle 1 (each cycle is 28 days)
  Defines as area under the plasma concentration versus time curve from time zero to the 24-hour sampling time.
[Stage 1 and Stage 2] PK parameters: area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC0-t) of HS-10352 | Cycle 1 Day 1 (C1D1)，at the first day of Cycle 1 (each cycle is 28 days)
  Defines as area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ).
[Stage 1] PK parameters: area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC0-t) of fulvestrant | From Cycle 1 to Cycle 2， each cycle is 28 days
  Defines as area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ).
[Stage 1 and Stage 2] PK parameters: the maximum concentration at steady-state (Css,max) of HS-10352 | Cycle 2 Day 1 (C2D1)，at the first day of Cycle 2 (each cycle is 28 days) each cycle is 28 days
  Defines as the maximum plasma drug concentration of HS-10352 at steady-state
[Stage 1] PK parameters: the maximum concentration at steady-state (Css,max) of fulvestrant | Cycle 2 (28 days)
  Defines as the maximum plasma drug concentration of fulvestrant at steady-state
[Stage 1 and Stage 2] PK parameters: time of the maximum concentration at steady state (Tss,max) of HS-10352 | Cycle 2 Day 1 (C2D1)，at the first day of Cycle 1 (each cycle is 28 days)
  Defined as the time to reach maximum plasma concentration following drug administration of HS-10352 at steady-state
[Stage 1] PK parameters: time of the maximum concentration at steady state (Tss,max) of fulvestrant | Cycle 2 (28 days)
  Defined as the time to reach maximum plasma concentration following drug administration of fulvestrant at steady-state
[Stage 1 and Stage 2] PK parameters: the minimum concentration at steady-state (Css,min) of HS-10352 | Cycle 2 Day 1 (C2D1)，at the first day of Cycle 1 (each cycle is 28 days)
  Defines as the minimum plasma drug concentration of HS-10352 at steady-state
[Stage 1 and Stage 2] PK parameters: the minimum concentration at steady-state (Css,min) of fulvestrant | Cycle 2 (28 days)
  Defines as the minimum plasma drug concentration of fulvestrant at steady-state
[Stage 1] Efficacy of HS-10352 in combination with fulvestrant: ORR | From the date of first dose until the date of disease progression or withdrawal from study, approximately 3 years
  ORR is defined as the proportion of participants with BOR of confirmed CR or confirmed PR based on assessment per RECIST v1.1.
[Stage 1 and Stage 2] Efficacy of HS-10352 in combination with fulvestrant: disease control rate (DCR) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 3 years
  The disease control was deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 6 weeks).
[Stage 1 and Stage 2] Efficacy of HS-10352 in combination with fulvestrant: duration of response (DoR) | From the date of CR, PR until the date of disease progression or withdrawal from study, approximately 3 years
  DOR only applies to participants whose best overall response is CR or PR based on assessment per RECIST v1.1. The start date is the date of first documented response of CR or PR (i.e. the start date of observed response, not the date when response was confirmed), and the end date is defined as the date of the first documented progression or death due to underlying cancer.
[Stage 1 and Stage 2] Efficacy of HS-10352 in combination with fulvestrant: progression free survival (PFS) | From the date of randomization or first dose (if randomization is not needed) until the date of disease progression or withdrawal from study, approximately 3 years
  PFS is defined as the time from the date of randomization or first dose (if randomization is not needed) to the date of the first documented progression or death due to any cause. PFS will be assessed per RECIST v1.1.
[Stage 2] Efficacy of HS-10352 in combination with fulvestrant: overall survival (OS) | From the date of randomization or first dose (if randomization is not needed) until the documentation of death from any cause, approximately 6 years
  OS is defined as the time from the date of randomization or first dose (if randomization is not needed) to the date of death due to any cause. For each participant who is not known to have died as of the cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China